CLINICAL TRIAL: NCT01331356
Title: Prospective Multicenter Pilot Study Evaluating the Analgesic Effect of an Injection of Botulinum Toxin Type A in the Ganglion Impar in Patients With Chronic Proctalgia According to the Criteria of Rome III
Brief Title: Analgesic Effect of an Injection of Botulinum Toxin Type A in the Ganglion Impar in Patients With Chronic Proctalgia
Acronym: Impartox
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10/4-T
Record Dates: First submitted 2011-03-31; First posted 2011-04-08 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-10

CONDITIONS: Proctalgia
Keywords: Chronic proctalgia; Botulinum toxin type A; Ganglion Impar; Perineal pain; Pudendal neuralgia; Refractory chronic proctalgia
MeSH Terms: conditions — Pudendal Neuralgia | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Injection of botulinum toxin type A (Experimental)
  Interventions: Drug: Botox

INTERVENTIONS:
Drug: Botox — One injection of botulinum toxin type A in the ganglion Impar in patients with chronic proctalgia

SUMMARY:
The main objective is to evaluate the analgesic efficacy of botulinum toxin type A in refractory chronic proctalgia one month after a bilateral injection of 50 units of Botox ® in the ganglion Impar (total dose = 100 units)

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient with chronic proctalgia according to the criteria of Rome III
* Chronic or recurrent rectal pain
* Pains evolve over periods of at least 20 minutes
* With the exclusion of other causes of rectal pain: ischemic, inflammatory bowel disease, cryptic lesions, intramuscular abscess, anal fissure, hemorrhoids, prostatitis and isolated coccydynia
* Pains evolve in a regular way since more than 3 months and the symptoms started since at least 6 months
* These chronic proctalgia include syndromes of anus elevator and nonspecific functional anorectal pains
* Patient with positive anesthetic block of ganglion Impar (minimum of 30 days before D0 and maximum of 270 days before D0)
* Main score (SP) ≥ 4 before infiltration of botulinum toxin type A
* Signed informed consent
* Subjects affiliated with an appropriate social security system

Exclusion Criteria:

* Pain related malignancy
* Patients with bleeding risk and recent anticoagulant therapy
* Surgery within 3 months
* Pre-existing anal incontinence
* Intolerance of botulinum toxin A, local anesthetics and radio contrast medium
* Injection of botulinum toxin in any place whatsoever in the previous 3 months
* Pregnancy and breast feeding
* Antibiotic treatment by aminoglycosides
* Recent anti-inflammatory treatment
* Severe myasthenia
* Lambert-Eaton syndrome
* Patients with neurological disorders, dysphagia, food choking or inhalation pneumonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in main score (SP) at 1 month | one month
  The main objective is to evaluate the analgesic efficacy of botulinum toxin type A in refractory chronic proctalgia one month after a bilateral injection of 50 units of Botox ® in the ganglion Impar (total dose = 100 units) by calculating the main score (SP).

SECONDARY OUTCOMES:
To assess the adverse events | 6 month
To assess the duration of action of the product (main score SP) | 6 month
To assess the changing parameters of quality of life: global improvement score / treatment satisfaction assessed by digital scale, international pain scales (MPI, QDSA, QCD) / Beck score and Hospital Anxiety and Depression (HAD) score | 6 month
To assess the evolution of analgesics consumption | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques LABAT, Dr, Principal Investigator — Nantes University Hospital
Locations (2):
- France (2):
  - Nantes University Hospital, Nantes
  - Centre Catherine de Sienne, Nantes